CLINICAL TRIAL: NCT07033130
Title: Early Feasibility, Exploratory, Within-subject, Acute Study Comparing the Performance of Different Sound Paths in Adult NeuroZti CI-users
Brief Title: The Performance of Different Sound Paths in Adult NeuroZti CI-users
Acronym: Percepolis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI5859
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06

CONDITIONS: Cochlear Implant; Hearing Loss, Bilateral or Unilateral
Keywords: cochlear implant; sound coding strategy; sound processor; speech perception; subjective measures
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sound paths in NeuroZti cochlear implant users (Experimental): NeuroZti cochlear implant users will complete speech perception testing and rate comfort and satisfaction between the Nuc8 and Neu2 sound paths.
  Interventions: Device: OMRP R2 + Percepolis Accessory Software; Device: Nuc8 Sound Path; Device: Neu2 Sound Path

INTERVENTIONS:
Device: OMRP R2 + Percepolis Accessory Software — The Oticon Medical Research Platform Release 2 (OMRP R2) + Percepolis Accessory Software is an investigational or research tool that includes hardware, firmware and software elements, which can connect to an Oticon Medical Cochlear Implant (CI). It is intended to be used exclusively for research with Oticon Medical CI users participating in research experiments or clinical studies. The hardware components are referred to as 'OMRP R2' and the software components are called 'Percepolis Accessory Software'.
Device: Nuc8 Sound Path — Nuc8 is the sound path used in Cochlear Nucleus Sound Processors.
Device: Neu2 Sound Path — Neu2 is the sound path that is currently used in the Neuro 2 Sound Processor.

SUMMARY:
The goal of this clinical trial is to compare speech perception and user satisfaction between two sound paths, Nuc8 (Cochlear Nucleus sound path) and Neu2 (Neuro 2 sound path), in adult users of the NeuroZti cochlear implant.

Following Cochlear's acquisition of Neurelec, there is a need to support existing NeuroZti implant users who currently rely on the Neuro 2 sound processor. The Nuc8-based sound processor, currently in development, is designed to be compatible with the Neuro system while integrating with Cochlear's ecosystem of tools and applications developed over the past decade.

To ensure long-term support and maintainability, transitioning to the Nuc8 sound path is preferred. However, changes in sound paths may impact sound quality, speech perception, and user acceptance.

The main question this study aims to answer is: how does speech performance and user satisfaction compare between the Nuc8 and Neu2 sound paths?

Participants will:

* Undergo speech perception testing in quiet environments
* Provide ratings on comfort and overall satisfaction

The study involves a single visit lasting approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old at time of consent.
2. Post-lingually deafened.
3. Bilaterally or unilaterally implanted with Oticon Medical Neuro ZTI cochlear implant, using Crystalis with autoXDP (GMCI 'CAP') as the main program, at 500pps stimulation rate. For bilateral CI users, only first-implanted side will be tested.
4. Fluent in French as determined by the investigator.
5. Willing to participate and comply with requirements of the protocol
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Additional health complexities that would prevent or restrict participation in the evaluations, including significant visual impairment and/or cognitive impairment.
2. Subjects who have life sustaining devices (such as pacemakers).
3. NeuroZti Subjects with Antenna SD Type.
4. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
5. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
6. Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
7. Pregnant or breastfeeding women.
8. Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by investigator or Sponsor to not impact this investigation).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage disyllabic word recognition Fournier scores in quiet at stimulated input level of 65 dB SPL for both Nuc8 and Neu2 sound paths | Day 0 (Study Visit 1)
  This involves testing open-set speech perception performance at simulated input of 65 dB SPL, which represents speech spoken at a normal conversational level. The word test will be performed in the sound field at 0° azimuth. Upon hearing the word, participants are instructed to repeat back the word, and the experimenter will score the recognition correct as either correct (i.e., when the subject repeat the exact word) or incorrect (i.e., when the subject does not repeat the exact word).

SECONDARY OUTCOMES:
Percentage disyllabic word recognition scores in quiet at stimulated input level of 55 dB SPL and at 40 dB SPL for both Nuc8 and Neu2 sound paths | Day 0 (Study Visit 1)
  This involves testing softer levels of 55 dB SPL and 40 dB SPL to investigate differences in speech coding and dynamic range management system over a range of levels.
Occurrence rate of preference using Neu2 and Nuc8 configurations for four subjective preference questions | Day 0 (Study Visit 1)
  This outcome measure involves a comparison of subjective comfort and satisfaction with Neu2 versus Nuc8 sound paths. Participants will judge the quality and comfort of various sounds that are presented, answering four questions:
  Q1: Which one sounds louder? Q2: Which one sounds clearer? Q3: Which one sounds more pleasant? Q4: Which one do you prefer listening to everyday in your behind the ear sound processor?

CONTACTS AND LOCATIONS:
Overall Officials: PRS Specialist, Study Director — Cochlear
Locations (1):
- Cochlear Vallauris, Vallauris, France

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.